CLINICAL TRIAL: NCT00928980
Title: The Clinical and Cost-effectiveness of Mindfulness Based Cognitive Therapy, Maintenance Antidepressant Medication and Its Combination in the Prevention of Relapse in Patients With Recurrent Depression
Brief Title: Mindfulness Based Cognitive Therapy and Antidepressant Medication in Recurrent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Anne Speckens, Prof. dr. Anne E.M. Speckens, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFN-2009-2013; 80-82310-98-09018; 2008/242
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Depressive Disorder, Major
Keywords: Recurrent Major Depressive Disorder; Mindfulness Based Cognitive Therapy; Cost-effectiveness; Antidepressant medication; Randomized Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness Based Cognitive Therapy and withdrawal of antidepressant medication between the 4th and 5th session, patients being off medication until the end of study period (15 months).
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Combination (Experimental): Mindfulness Based Cognitive Therapy combined with the use of antidepressant medication during the study (15 months).
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy; Drug: Optimal Medical Care
- Optimal Medical Care (Active Comparator): Treatment with optimal medical care: therapeutic dose of antidepressant medication during at least 15 months, administered in accordance with current guidelines.
  Interventions: Drug: Optimal Medical Care

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Mindfulness Based Cognitive Therapy is an 8-week during group intervention encompassing meditation practice and cognitive therapy techniques.
  Arms: Combination; Mindfulness Based Cognitive Therapy
Drug: Optimal Medical Care — Therapeutic dose of antidepressant medication
  Arms: Combination; Optimal Medical Care

SUMMARY:
The purpose of this study is to investigate the (cost)effectiveness of mindfulness based cognitive therapy (MBCT) compared to that of antidepressant medication, and its combination with regard to the prevention of relapse or recurrence in patients with recurrent depression.

DETAILED DESCRIPTION:
In the Netherlands, treatment as usual for patients with (recurrent) Major Depressive Disorder consists of maintenance antidepressant medication. Mindfulness-based cognitive therapy (MBCT) is a recently developed psychological intervention that appears to be promising in terms of preventing relapse or recurrence in patients with recurrent depression. It consists of 8 weekly group sessions in which meditation exercises are combined with cognitive therapeutic elements such as identifying negative thoughts and monitoring and scheduling activities.

In this study, the (cost)effectiveness of a) MBCT on its own, b) antidepressant medication on its own and c) the combination of MBCT and antidepressant medication will be investigated in 350 patients with recurrent depression who are currently in remission.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent Major Depressive Episode (at least 3 previous episodes)
* Treatment with therapeutic dose of antidepressant medication during past six months
* Currently in full or partial remission

Exclusion Criteria:

* Bipolar disorder (current and previous (hypo)manic episodes)
* Psychotic disorder (current and previous)
* Neurological or somatic illness affecting depression or outcome measures
* Current alcohol or drugs dependency
* Use of high dosage benzodiazepines (> 2 mg Lorazepam equivalents daily)
* Recent Electro Convulsive Therapy (< 3 months ago)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relapse/recurrence of Major Depressive Episode | 3, 6, 9, 12, 15 months
  Relapse or recurrence of depression will be assessed trimonthly using the Structured Clinical Interview for DSM-V (SCID) depression module.

SECONDARY OUTCOMES:
Costs made by consumption of medical care and production loss | 3, 6, 9, 12, 15 months
  Using prospective calendars and retrospective questionnaires about contacts with health care in the past 3 months (assessed trimonthly) we will estimate the costs of depression health care and the quality of life (selfreport). We will compare the cost-effectiveness ratios between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (13):
- Netherlands (13):
  - Pro Persona, Arnhem, Gelderland
  - Pro Persona, Ede, Gelderland
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Pro Persona, Tiel, Gelderland
  - GGZ Noord-Holland-Noord, Alkmaar, North Holland
  - Free University Medical Center and GGZ In Geest, Amsterdam, North Holland
  - AMC Amsterdam, Amsterdam, North Holland
  - GGZ Rivierduinen - Leiden, Leiden, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - PsyQ, The Hague, South Holland
  - Parnassia ACO Zuid, The Hague, South Holland
  - GGZ Centraal, Amersfoort, Utrecht
  - GGZ Duin- en Bollenstreek, Katwijk

REFERENCES:
- [Background] Kuyken W, Byford S, Taylor RS, Watkins E, Holden E, White K, Barrett B, Byng R, Evans A, Mullan E, Teasdale JD. Mindfulness-based cognitive therapy to prevent relapse in recurrent depression. J Consult Clin Psychol. 2008 Dec;76(6):966-78. doi: 10.1037/a0013786. PMID 19045965
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Derived] Huijbers MJ, Wentink C, Simons E, Spijker J, Speckens A. Discontinuing antidepressant medication after mindfulness-based cognitive therapy: a mixed-methods study exploring predictors and outcomes of different discontinuation trajectories, and its facilitators and barriers. BMJ Open. 2020 Nov 11;10(11):e039053. doi: 10.1136/bmjopen-2020-039053. PMID 33177138
- [Derived] Huijbers MJ, Spinhoven P, Spijker J, Ruhe HG, van Schaik DJ, van Oppen P, Nolen WA, Ormel J, Kuyken W, van der Wilt GJ, Blom MB, Schene AH, Rogier A, Donders T, Speckens AE. Discontinuation of antidepressant medication after mindfulness-based cognitive therapy for recurrent depression: randomised controlled non-inferiority trial. Br J Psychiatry. 2016 Apr;208(4):366-73. doi: 10.1192/bjp.bp.115.168971. Epub 2016 Feb 18. PMID 26892847
- [Derived] Huijbers MJ, Spinhoven P, Spijker J, Ruhe HG, van Schaik DJ, van Oppen P, Nolen WA, Ormel J, Kuyken W, van der Wilt GJ, Blom MB, Schene AH, Donders AR, Speckens AE. Adding mindfulness-based cognitive therapy to maintenance antidepressant medication for prevention of relapse/recurrence in major depressive disorder: Randomised controlled trial. J Affect Disord. 2015 Nov 15;187:54-61. doi: 10.1016/j.jad.2015.08.023. Epub 2015 Aug 18. PMID 26318271
- [Derived] Huijbers MJ, Spijker J, Donders AR, van Schaik DJ, van Oppen P, Ruhe HG, Blom MB, Nolen WA, Ormel J, van der Wilt GJ, Kuyken W, Spinhoven P, Speckens AE. Preventing relapse in recurrent depression using mindfulness-based cognitive therapy, antidepressant medication or the combination: trial design and protocol of the MOMENT study. BMC Psychiatry. 2012 Aug 27;12:125. doi: 10.1186/1471-244X-12-125. PMID 22925198